CLINICAL TRIAL: NCT00008424
Title: A Phase I Study of Irinotecan in Patients With Refractory Solid Tumors Who Are Concomitantly Receiving Anticonvulsants
Brief Title: Irinotecan in Treating Children With Refractory or Advanced Solid Tumors Who Are Receiving Anticonvulsants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: P9871; COG-P9871 (Other: Children's Oncology Group); POG-P9871 (Other: Pediatric Oncology Group); CDR0000068410 (Other: Clinicaltrials.gov)
Record Dates: First submitted 2001-01-06; First posted 2003-06-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of irinotecan in treating children with refractory or advanced solid tumors who are receiving anticonvulsants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of irinotecan in children with refractory or advanced solid tumors receiving anticonvulsants.
* Determine the dose-limiting toxicity of irinotecan in this patient population.
* Evaluate the pharmacokinetic behavior of this treatment regimen in these patients.
* Determine, preliminarily, the antitumor activity of this treatment regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to type of concurrent anticonvulsant (enzyme activating anticonvulsants vs valproic acid vs other anticonvulsants).

Patients receive irinotecan IV over 1 hour daily for 5 days. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 6 months for up to 4 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 3-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy refractory to conventional therapy or for which no conventional therapy exists

  * Histologic confirmation not required for brain stem tumors
* Concurrently on anticonvulsants at a steady level for at least 2 weeks

PATIENT CHARACTERISTICS:

Age:

* 1-21 years old

Performance status:

* Karnofsky 50-100% (over 10 years of age)
* Lansky 50-100% (10 years of age or under)

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Neutrophil count at least 1,000/mm3
* Platelet count at least 100,000/mm3 (transfusion independent)
* Hemoglobin at least 8.0 g/dL (red blood cell transfusions allowed)

Hepatic:

* Bilirubin no greater than 1.5 times normal for age
* SGPT less than 5 times normal for age
* Albumin at least 2 g/dL

Renal:

* Creatinine no greater than 1.5 times normal for age OR
* Creatinine clearance or radioisotope glomerular filtration rate at least lower limit of normal for age

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No evidence of active graft-vs-host disease
* Neurologic deficits for CNS tumors stable for at least 2 weeks prior to study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 1 week since prior antineoplastic biologic therapy
* At least 6 months since prior allogeneic stem cell transplantation
* At least 1 week since prior growth factors
* No concurrent sargramostim (GM-CSF)
* No concurrent prophylactic growth factors during first course of study therapy
* Recovered from prior immunotherapy

Chemotherapy:

* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosourea) and recovered

Endocrine therapy:

* Concurrent dexamethasone for CNS tumors with increased intracranial pressure allowed if dose stable or decreasing for at least 2 weeks prior to study

Radiotherapy:

* At least 2 weeks since prior local palliative radiotherapy (small part)
* At least 6 months since prior craniospinal radiotherapy
* At least 6 months since prior radiotherapy to at least 50% of pelvis
* At least 6 weeks since prior substantial bone marrow radiotherapy
* Recovered from prior radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational agent

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2000-10; Primary Completion 2005-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose (MTD) of irinotecan

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moghrabi, MD, Study Chair — Hopital Sainte Justine
Locations (51):
- United States (45):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Children's Hospital of Denver, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Floating Hospital Infants and Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - CCOP - Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec